CLINICAL TRIAL: NCT01179698
Title: Navigation Surgery for Bone and Soft Tissue Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sungwook Seo, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-08-058
Record Dates: First submitted 2010-07-30; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Bone Tumors
Keywords: computer-assisted surgery; bone tumor; We will evaluate whether computer-assisted surgery; will be feasible and safe for bone tumor resection
MeSH Terms: conditions — Bone Neoplasms | interventions — Surgery, Computer-Assisted; Surgical Navigation Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stryker navigation system (Other)
  Interventions: Procedure: Navigation surgery; Procedure: Navigation system

INTERVENTIONS:
Procedure: Navigation surgery — In en bloc resection, the osteotomy sites were determined by navigation guidance. For curettage, we monitored curette in real-time with navigation.
Procedure: Navigation system — In en bloc resection, the osteotomy sites were determined by navigation guidance. For curettage, we monitored curette in real-time with navigation.

SUMMARY:
Bone tumor near the articular cartilage is hard to remove sufficiently without damaging adjacent joint. The purpose of this study was to evaluate the feasibility of navigation-assisted surgery for saving joint in bone tumor resection or curettage. In this study, the investigators hypothesized that computer-assisted surgery is feasible method to get both enough margin and joint salvage. Each of them is important intermediate factor for either oncologic outcome or functional outcome respectively. The investigators designed this study to find what proportion of patients who underwent computer-assisted resection could get enough margins using some criteria obtained by overlapping preoperative and postoperative images. The investigators also evaluated whether computer-assisted surgery can be feasible for joint saving using some criteria including functional outcome.

ELIGIBILITY:
Inclusion criteria:

1. First condition is that the benign tumor is located deeply in bones of extremities, or pelvis, so we anticipate the difficulty to find the tumor and to assess the adequacy of resection without the aid of computer-assisted navigation during operation.
2. Second condition is when the violation of joint or growth plate is expected during removal of tumor due to its close proximity to joint or growth plate.

In case of malignant bone tumor, the sufficient preservation of joint anatomy should be required even with resection margin of 1.5 cm away from reactive zone of tumor. The sufficient preservation of joint is defined when at least 1 cm subchondral bone is remained after tumor resection, because 1 cm subchondral bone is required for fixation with allograft in subsequent reconstruction. The sufficient preservation of joint is also defined when articular surface is removed, but more than 50% of articular surface has to be saved.

Exclusion criteria were

1. Patients who denied to perform navigation surgery after explanation of navigation surgery protocol
2. Medically high-risk patients who could not withstand long surgical time for joint reconstruction
3. Patients whose feasibility of joint preservation was not fulfill the above inclusion criteria at initial presentation, although the tumor size was decreased enough to fulfill the inclusion criteria in MRI after completion of neoadjuvant chemotherapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Resection margin and safety | Day 1 - During operation
  Pre-operative and post-operative CT or MRI images were fused using image fusion application of navigation software (Striker, Mahwah, NJ)in order to evaluate the resection margin.
Resection margin and safety | 3 months - postoperative
  Pre-operative and post-operative CT or MRI images were fused using image fusion application of navigation software (Striker, Mahwah, NJ)in order to evaluate the resection margin.

SECONDARY OUTCOMES:
Oncological outcome and functional score | Postoperative 6 month and 12month
  1) Oncological outcome after 6 month or 12 month from surgery like patient survival or tumor recurrence (tumor recurrence was diagnosed with PET CT or MRI according to the nature of original tumor), 2) functional scores were assessed by evaluation systems of the Musculoskeletal Tumor Society (MSTS)and Toronto Extremity Salvage Score (TESS).

CONTACTS AND LOCATIONS:
Overall Officials: Sung Wook Seo, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Irwon-Dong, South Korea